CLINICAL TRIAL: NCT04902157
Title: Relationship Between CT- Value With Prognosis in COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, nooshin dalili, assistant Professor of SBMU, Shahid Beheshti University of Medical Sciences
Other Study IDs: SBMU.34.675
Record Dates: First submitted 2021-05-25; First posted 2021-05-26 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cycle threshold — cycle threshold number

SUMMARY:
evaluate the relationship between cycle threshold number with final prognosis in COVID-19 patients

DETAILED DESCRIPTION:
evaluate the relationship between cycle threshold number with final prognosis in COVID-19 patients

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 PCR positive

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 PCR Positive
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
prognosis | 6 months
  death or alive

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - SBMU, Tehran
  - Nooshin Dalili, Tehran

IPD SHARING:
Plan to Share IPD: No